CLINICAL TRIAL: NCT06225024
Title: Evaluation of the Efficacy of Extracorporeal Shock Wave Therapy (ESWT) Following Botulinum Toxin Type A Injection on Post-Stroke Ankle Plantar Flexor Spasticity
Brief Title: Efficacy of Extracorporeal Shock Wave Therapy on Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Havva Talay Çalış, Prof, Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Health Sciences
Record Dates: First submitted 2024-01-07; First posted 2024-01-25 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Spasticity, Muscle
Keywords: Botulinum Toxin A; ESWT; Stroke; Spasticity; Modified Ashworth Scale; Heckmatt Scale
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Cardiac Resynchronization Therapy Devices; incobotulinumtoxinA; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled
Who Masked: Outcomes Assessor
Masking Description: The patients in both groups underwent the following evaluations before treatment, at one month and three months after treatment by a treatment-blinded Physical Medicine and Rehabilitation (PMR) physician:
  1. Modified Ashworth Scale (MAS)
  2. Brunnstrom Motor Recovery Stage (BMRS)
  3. Ankle range of motion (2) measurement
  4. Clonus score (CS)
  5. Barthel Index (BI)
  6. Heckmatt measurements with ultrasonography
  7. Visual analog scale (VAS) pain assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BoNT-A (Active Comparator): BoNT-A was injected into the affected gastrocnemius muscle under ultrasonography guidance at doses recommended by standard guidelines and appropriate for the patient (50 IU to the medial head, 25 IU to the lateral head). In addition, conventional physical therapy exercises (stretching exercises, range of motion (ROM) exercises, neurophysiologic exercises, and gait exercises) were applied to the patients five days a week for four weeks.
  Interventions: Drug: BoNT A
- BoNT-A and ESWT (Experimental): In addition to the treatments (BoNT-A injection and exercise) in Group 1, one week after the injection, a total of 4 sessions (2 days a week) of ESWT (1000 impulses with an energy density of 0.1 mj/mm2, pressure of 2 bar, and frequency of 4 Hz) were applied to the medial and lateral heads of the gastrocnemius muscle.
  Interventions: Device: ESWT; Drug: BoNT A

INTERVENTIONS:
Device: ESWT — Extracorporeal shock wave therapy (ESWT) is a treatment method based on high-intensity sound waves focusing on the desired body area to provide treatment. ESWT is a safe, non-invasive, alternative treatment for spasticity in patients with stroke, cerebral palsy, and multiple sclerosis and does not cause muscle weakness or adverse effects
  Other Names: device therapy
  Arms: BoNT-A and ESWT
Drug: BoNT A — BoNT-A is widely recognized as the benchmark for enhancing the effectiveness of spasticity management
  Other Names: drug therapy

SUMMARY:
Introduction: We aimed to compare the efficacy of Botulinum Toxin Type A(BoNT-A) injection and BoNT-A injection in combination with ESWT for post-stroke lower extremity ankle plantar flexor spasticity.

Materials and Method: Patients with post-stroke ankle plantar flexor spasticity of 1 or more on the modified Ashworth Scale(MAS) were randomized into two groups.

Group 1(n:20): BoNT-A was injected into the gastrocnemius muscle and conventional physical therapy exercises were performed.

Group 2(n:20): ESWT was applied to the gastrocnemius muscle in addition to the treatments in group 1.

DETAILED DESCRIPTION:
Group 1 (n:20): BoNT-A was injected into the affected gastrocnemius muscle under ultrasonography guidance at doses recommended by standard guidelines and appropriate for the patient (50 IU to the medial head, 25 IU to the lateral head). In addition, conventional physical therapy exercises (stretching exercises, range of motion (ROM) exercises, neurophysiologic exercises, and gait exercises) were applied to the patients five days a week for four weeks.

Group 2 (n:20): In addition to the treatments (BoNT-A injection and exercise) in Group 1, one week after the injection, a total of 4 sessions (2 days a week) of ESWT (1000 impulses with an energy density of 0.1 mj/mm2, pressure of 2 bar, and frequency of 4 Hz) were applied to the medial and lateral heads of the gastrocnemius muscle.

The patients in both groups underwent the following evaluations before treatment, at one month and three months after treatment by a treatment-blinded Physical Medicine and Rehabilitation (PMR) physician.

Patients' age, sex, occupation, hemiplegic sides, and etiology of hemiplegia were recorded. Physical examination was performed, and examination findings were recorded. The presence of post-treatment pain, redness, tenderness, or other adverse findings were questioned.

MAS, Brunnstrom Motor Recovery Stage(BMRS), ankle range of motion(ROM) measurement, clonus score(CS), Barthel Index(BI), Heckmatt measurements with ultrasonography, and visual analog scale(VAS) evaluations were performed on the patients.

ELIGIBILITY:
Inclusion criteria:

* Being diagnosed with stroke according to the definition of the World Health Organization in 1989
* Having a stroke confirmed by computed tomography (CT) and magnetic resonance imaging (MRI)
* Being aged over 18 years
* Having a MAS score of 1 and above for gastrocnemius, the plantar flexor muscle of the ankle
* Having a stable general condition after a stroke
* Giving consent to participate in the study.

Exclusion criteria:

* Having a fixed contracture in the ankle
* Having no spasticity in the soleus, the plantar flexor muscle of the ankle
* Previous antispastic surgery performed on the area
* Change in antispastic drug use in the last six months, if any
* Injection of BoNT-A, alcohol, phenol, or any other substance into the area in the last six months
* Active infection or cancer at the application site
* Having a cardiac pacemaker
* Having bleeding diathesis
* Having vascular complaints such as deep vein thrombosis, venous stasis, phlebitis, arterial disease
* Being pregnant
* Having neuromuscular junction disease or motor neuron disease
* Having a known allergy to BoNT-A
* 12. Active use of aminoglycosides or other antibiotic groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | at baseline, at one month and three months after treatment
  This scale is used to evaluate the severity of spasticity. MAS is based on a subjective evaluation of the resistance felt during the examination.
  0: No tone increase
  1. Slight increase in tone characterized by a catch and release or minimal resistance at the end of the range of motion 1+: Slight increase in muscle tone with minimal resistance throughout less than half of the range of motion
  2. Increased muscle tone throughout the entire range of motion, but joints can be easily moved
  3. Considerable increase in tone; passive movement is difficult
  4. Affected parts are rigid in flexion and extension.

SECONDARY OUTCOMES:
Brunnstrom Motor Recovery Stage (BMRS) | at baseline, at one month and three months after treatment
  It is a motor function assessment scale to evaluate the motor development of hemiplegic patients. According to Brunnstrom, there are six stages in the recovery process of hemiplegic patients, and the upper extremity, lower extremity, and hands are individually evaluated. A higher BMRS indicates better motor development

OTHER OUTCOMES:
Ankle ROM measurement | at baseline, at one month and three months after treatment
  Passive joint ROM of the affected ankle was calculated using a goniometer according to the neutral zero method.
Clonus score (CS) | at baseline, at one month and three months after treatment
  The clonus felt during the examination is graded from 0 to 3. The study evaluated the clonus score by grading the clonus felt while passively moving the affected ankle from maximum plantar flexion to maximum dorsiflexion.
  The clonus scores were interpreted as 0= None, 1= Non-sustained, 2= Sustained, and 3=Spontaneous/Light touch-induced.
Barthel Index (BI) | at baseline, at one month and three months after treatment
  BI is a detailed, objective, easy-to-administer, and comprehensible scale that assesses physical independence in activities of daily living and thoroughly evaluates all steps of activities of daily living. It was developed to assess the change in functional status in rehabilitation patients. BI consists of 10 main topics. Feeding, transfers from bed to wheelchair and back, grooming, toileting, bathing, mobility on level surfaces (using a wheelchair if appropriate), climbing up and downstairs, dressing, bowel care, and bladder care are questioned. A score of 0-20 indicates complete dependence; a score of 21-61 indicates severe dependence; a score of 62-90 indicates moderate dependence; a score of 91-99 indicates mild dependence; a score of 100 indicates complete independence.
Heckmatt measurements with ultrasonography | at baseline, at one month and three months after treatment
  The echo intensity within the affected muscle group is assessed and scored with the help of ultrasonography. Echo intensity in the gastrocnemius muscle was visually evaluated in transverse view using a linear probe (Philips Clearvue 550) with an imaging frequency of 5-12 MHz in sonographic examination according to the Heckmatt scale; grade I was recorded as normal; grade II as increased muscle echo intensity with considerable bone echo; grade III as a significant increase in muscle echo intensity and decreased bone echo; grade IV as very high muscle echo intensity and complete loss of bone echo.
Visual analog scale (VAS) pain assessment. | at baseline, at one month and three months after treatment
  A 10-centimeter line was drawn for pain, one end indicates no pain, and the other indicates severe pain. The patient was asked to mark his/her current condition on this line. The length of the distance from the end which indicates no pain to the point where the patient marks indicates the patient's pain

CONTACTS AND LOCATIONS:
Overall Officials: HAVVA TALAY ÇALIŞ, Principal Investigator — KAYSERİ CITY HOSPITAL
Locations (1):
- Health Sciences University, Kayseri Medicine Faculty, Kayseri, Kocasinan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoldas Aslan S, Kutlay S, Dusunceli Atman E, Elhan AH, Gok H, Kucukdeveci AA. Does extracorporeal shock wave therapy decrease spasticity of ankle plantar flexor muscles in patients with stroke: A randomized controlled trial. Clin Rehabil. 2021 Oct;35(10):1442-1453. doi: 10.1177/02692155211011320. Epub 2021 Apr 28. PMID 33906450
- [Background] Yang E, Lew HL, Ozcakar L, Wu CH. Recent Advances in the Treatment of Spasticity: Extracorporeal Shock Wave Therapy. J Clin Med. 2021 Oct 14;10(20):4723. doi: 10.3390/jcm10204723. PMID 34682846